CLINICAL TRIAL: NCT02537249
Title: Effects of Dexmedetomidine on Quality of Recovery and Analgesia After Video-assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2015-0556
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer; Video-assisted Thoracoscopic Surgery
Keywords: dexmedetomidine; quality of recovery
MeSH Terms: conditions — Lung Neoplasms | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Saline 0.9% (Sham Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Formula for administrated were randomized by computer-generated randomization. The patients and anesthesiologist, who administered and conducted all this trial, were blinded to the medication allocation. An anesthesiologist, who responsible for preparation of medication was the only person, recognized of the randomization code during trial. After one-lung ventilation, dexmedetomidine group would start the loading of dexmedetomidine (1μg/kg) during 20 minutes.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Normal saline — Saline placebo infusion will be adjusted the same fashion as the active comparator drug.
  Other Names: Saline 0.9%
  Arms: Saline 0.9%

SUMMARY:
Dexmedetomidine is a selective α2 adrenergic agonist that can be considered analgesics, anxiolytic,and anti-stress effect . This randomized, double-blind placebo-controlled trial of intraoperative dexmedetomidine for improvement of quality of recovery and analgesia from surgery. Patients scheduled to undergo video-assisted thoracoscopic surgery (VATS) will be enrolled. Patients will be recruited before the date of their surgery and will complete the Quality of Recovery-40 (QoR-40) questionnaire before their surgery and at 24 and 48 hours post op. They will also complete clinically significant pains score and oxygenation from the postanesthetic recovery unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

1. The inclusion criteria included patients scheduled video-assisted thoracoscopic surgery for lung cancer
2. Adults above 20 years of age and providing informed consent.
3. American Society of Anesthesiologists (ASA) Physical class II, & III patients

Exclusion Criteria:

1. severe functional liver or kidney disease
2. history of chronic pain requiring opioid treatment
3. arrhythmia or received treatment with antiarrythmic drug .
4. severe bradycardia (HR < 45 bpm) and AV block
5. pathologic esophageal lesion (esophageal stricture or varix )
6. pregnancy
7. psychiatric/central nervous system disturbance that would preclude completion of the QoR-40 questionnaire
8. History of alcohol or drug abuse

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
quality of recovery measured by QoR-40 questionnaire | 24 hr after operation
pulmonary function test | 24 hr after operation
  postoperative lung function assessed by spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Seoul, South Korea